CLINICAL TRIAL: NCT05668572
Title: A Multi-centre, Blinded, Randomized and Gardasil-controlled Phase III Trial to Evaluate the Efficacy, Immunogenicity and Safety Profile of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli)
Brief Title: A Phase III Trial Evaluates the Efficacy, Immunogenicity and Safety Profile of HPV Vaccine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Health Guard Biotechnology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLWS-V502-03
Record Dates: First submitted 2022-12-06; First posted 2022-12-30 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Human Papillomavirus Infection
Keywords: CIN 2/3; AIS; Invasive Cervical Carcinoma; VIN 2/3; VaIN 2/3; Anal Intraepithelial Neoplas
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Sponsor, investigators and biostatisticians will remain blinded to subject allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Group of Investigational Vaccine (Experimental)
  Interventions: Biological: Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli)
- The Group of Active Control Vaccine (Active Comparator)
  Interventions: Biological: Recombinant Quadrivalent Human Papillomavirus (Types 6,11,16,18) Vaccine (Saccharomyces cerevisiae)（GARDASIL®）

INTERVENTIONS:
Biological: Recombinant Nonavalent (types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia coli) — 0.5-mL suspension for injection, each 0.5-mL prefilled syringe dose contains L1 proteins of HPV types 6/11/16/18/31/33/45/52/58 in the amounts of 30mcg, 40mcg, 60mcg, 40mcg, 20mcg, 20mcg, 20mcg, 20mcg and 20mcg, respectively, totaling 270mcg of antigens. A 3-dose regimen administered at months 0, 2 and 6.
  Arms: The Group of Investigational Vaccine
Biological: Recombinant Quadrivalent Human Papillomavirus (Types 6,11,16,18) Vaccine (Saccharomyces cerevisiae)（GARDASIL®） — 0.5-mL suspension for injection, each 0.5-mL single-dose syringe contains approximately 20 mcg of HPV Type 6 L1 protein, 40 mcg of HPV Type 11 L1 protein, 40 mcg of HPV Type 16 L1 protein, 20 mcg of HPV Type 18 L1 protein, totaling 120 mcg of antigens
  Arms: The Group of Active Control Vaccine

SUMMARY:
This study is to demonstrate that the administration of the investigational vaccine can reduce the Combined Incidence of HPV types 6/11/16/18/31/33/45/52/58-related high-grade Cervical Intraepithelial Neoplasia (CIN 2/3), Adenocarcinoma in Situ (AIS), Invasive Cervical Carcinoma, high-grade Vulvar Intraepithelial Neoplasia (VIN 2/3), high-grade Vaginal Intraepithelial Neoplasia (VaIN 2/3), high-grade Anal Intraepithelial Neoplasia (AIN 2/3), vulvar cancer, vaginal cancer or anal cancer.

DETAILED DESCRIPTION:
This is a multi-center, blinded, randomized and Gardasil-controlled (quadrivalent HPV vaccine GARDASIL®) Phase III clinical study. The study will recruit a total of approximately 12,000 healthy Chinese women ages 20-45 years with permanent residence, who will be randomized at a 1: 1 ratio to receive the investigational vaccine or the positive control (quadrivalent HPV vaccine GARDASIL®), respectively.

Healthy women ages 20-45 eligible for the study will be stratified at a 2: 2: 1 ratio into three age subgroups (i.e. 20-26 years of age, 27-35 years of age and 36-45 years of age), and each subgroup will be randomized at a 1: 1 ratio to receive the investigational vaccine or the positive control (quadrivalent HPV vaccine GARDASIL®), respectively. A total of 1,000 subjects will be allocated to an Immunogenicity Cohort, who will also be randomized at a 1: 1 ratio to receive the investigational vaccine or the positive control. The Immunogenicity Cohort is set up to evaluate the immune responses induced by the investigational vaccine and their persistence.

For the Sample allocation plan, twelve thousand (12,000) subjects from the chosen clinical trial sites are stratified at a 2: 2: 1 ratio into 3 age subgroups, i.e. 4,800 in the subgroup of ages 20-26 years, 4,800 in the subgroup of ages 27-35 years, and 2,400 in the subgroup 36-45 years of age.

Immunogenicity evaluation will be conducted at a clinical trial site in 1,000 subjects, selected randomly in the order of enrollment.

The Primary study objectives also involve:

-To demonstrate that administration of the investigational vaccine reduces the Combined Incidence of HPV types 6/11/16/18/31/33/45/52/58-related persistent infections, and cervical, vulvar, vaginal and anal lesions detected in samples from three or more consecutive visits (+/-1 month visit window) 12 months or longer apart.

The Secondary study objectives involve:

* To evaluate the safety profile of the investigational vaccine in healthy women ages 20-45;
* To demonstrate that geometric mean titers of antibody responses specific to HPV types 6/11/16/18 induced by the investigational vaccine are non-inferior to those generated by GARDASIL;
* To demonstrate that the investigational vaccine produces antibody responses specific to HPV types 31/33/45/52/58;
* To evaluate the levels and persistence of antibody responses against HPV types 6/11/16/18/31/33/45/52/58 generated by the investigational vaccine;
* To demonstrate that the investigational vaccine reduces the Combined Incidence of HPV types 6/11/16/18/31/33/45/52/58-related persistent infections detected in samples from 2 or more consecutive visits 6 months (+/-1 month visit window) or longer apart.

The Exploratory study objectives involve:

* To evaluate the impact of a 3-dose regimen of the investigational vaccine on the incidence of HPV types 6/11/16/18/31/33/45/52/58-related cytological abnormalities (ASC-US, positive for high-risk HPV types, or worse) as determined by the Thinprep cytologic test (TCT test) among subjects, who are naïve (seronegative) to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain negative to the relevant HPV type(s) as determined by HPV-DNA test and without abnormal cervical biopsy result through Month 7;
* To evaluate the incidence of non-vaccine HPV type-related Cervical Intraepithelial Neoplasia (CIN), Adenocarcinoma in Situ (AIS) and Cervical Carcinoma as determined by histopathologic examination post 3 doses of the investigational vaccine;
* To evaluate the incidence of non-vaccine HPV type-related persistent infections for no less than 6 months, and cervical, vulvar, vaginal and anal diseases as determined by histopathologic examination post 3 doses of the investigational vaccine;
* To evaluate the incidence of non-vaccine HPV type-related cytological abnormalities (ASC-US, positive for high-risk HPV types, or worse) as determined by the TCT test post 3 doses of the investigational vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects ages ≥20 and <46 (i.e. 20-45 years of age).
* Subjects who voluntarily agree to participate in the trial by giving written informed consent, fully understand of study procedures and the risks associated with participating in the study, and are aware of alternative interventions are available for those who do not participate in the trial.
* Subjects who are able to read, understand, and complete the daily diary card.
* Subjects who are in a good physical health as decided by the investigator based on his/her medical history and physical checkup results.
* Subjects who have had sexual activity prior to enrollment.
* Subjects who have refrained from sexual activity (including anal, vaginal, or genital/genital contact whether same sex or opposite sex) and agree to refrain from douching/vaginal cleansing, and using vaginal medications or preparations for 48 hours prior to any visit that includes collection of study specimens.

Note: if a subject does not meet this inclusion criterion, the Day 0 visit (at enrollment) may be rescheduled for a time when such criterion can be met.

* Subjects who are not pregnant (with negative urine pregnancy test) and breastfeeding at enrollment, and do not plan for pregnancy in the following 7 months; who have used effective contraception with no failures for 2 calendar days prior to the Day 0 visit (at enrollment), at the same time understand and agree that from Day 0 through Month 7, she shall not have sexual intercourse with males without effective contraception [Effective contraception is defined as the use of a marketed, approved contraceptive product that includes oral contraceptives, contraceptive injections, sub-dermal contraceptive implants, slow-release systems, contraception-patches, intrauterine devices (IUD), sterilization, abstinence, male condoms, contraceptive diaphragms, cervical cap].
* Subjects with an axillary temperature of 37.0 ℃ or less at enrollment.

Exclusion Criteria:

* Subjects who have received a marketed HPV vaccine, or have participated in an HPV vaccine clinical trial other than this one, or plan to receive an HPV vaccine other than the investigational vaccine or positive control during this study.
* Subjects who have a history of cervical cancer, CIN2+, HPV infections or an abnormal cytology result.
* Subjects who have a history of HPV-related external genital lesions (e.g. VIN, VaIN and genital warts), external genital cancer or vaginal cancer.
* Subjects who have a history of pelvic radiotherapy.
* Subjects who have had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Subjects who have hypertension or diabetes mellitus despite being treated by medication.
* Subjects who have a history of severe allergic reaction (e.g. anaphylactic shock, laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, Arthus reaction, etc.) to any prior vaccination or medication that required medical intervention.
* Subjects who are currently immunocompromised or have been diagnosed as having a congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease, or other autoimmune conditions.
* Subjects who have had a splenectomy.
* Subjects who are receiving or have received in the year prior to enrollment the following immunosuppressive therapies: radiation therapy, cyclophosphamide, azathioprine, methotrexate, any chemotherapy, cyclosporin, leflunomide (Arava™), TNF-α antagonists, monocolonal antibody therapies, intravenous gamma globulin (IVIG), antilymphocyte sera, or other therapy known to interfere with immune responses to the interventions.
* Subjects who are currently receiving systemic steroid therapy, or have received 2 or more courses of high dose systemic corticosteroids lasting at least 1 week in duration in the year prior to enrollment, with the exception of those who use inhaled, nasal, or topical corticosteroids.
* Subjects who have received any immune globulin product or blood-derived product within the 3 months prior to the first vaccination, or plan to receive any such product during the Day 0 through Month 7 period of the study.
* Subjects who have received inactivated vaccines within 14 days prior to the first vaccination or have received replicating (live attenuated) vaccines within 28 days prior to the first vaccination.
* Subjects who have thrombocytopenia or other coagulation disorder that would contraindicate intramuscular injections.
* Subject who have donated blood within 1 week prior to the first vaccination, or intend to donate during the Day 0 through Month 7 period of the study.
* Subjects who are expecting to donate eggs during the Day 0 through Month 7 period of the study.
* Subjects who are concurrently enrolled in clinical studies of other investigational or unregistered drug or vaccine, or studies involving collection of cervical specimens.
* Subjects who are unlikely to adhere to the study procedures, keep appointments, or are planning to relocate during the study.
* Subjects who have had a fever (defined as an axillary temperature ≥38.0 ˚C) within 3 days prior to the first vaccination or any acute illness that required systemic antibiotic and antiviral treatment within 5 days prior to the first vaccination.
* Subjects who have acute genital infections (e.g. acute vaginitis, acute endometritis, acute salpingitis, acute oophoritis) or gross purulent cervicitis.
* Subjects who are having menses (specimen collection at enrollment should be rescheduled for at least 3 days post the last day of the menstrual period).
* Subjects who do not have an intact cervix uteri or have more than one cervix uteri.
* Subjects who have a history or current evidence of other circumstances which might confound the results of the study, or which suggest it is not in the best interest of the subject to participate, as per the judgement of the investigator.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12000 (Actual)
Dates: Start 2020-12-05 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2023-02-23 (Estimated)

PRIMARY OUTCOMES:
The combined incidence of HPV types 6/11/16/18/31/33/45/52/58-related high-grade diseases | Up to 60th month after full immunization
  The combined incidence of HPV types 6/11/16/18/31/33/45/52/58-related high-grade Cervical Intraepithelial Neoplasia (CIN 2/3), Adenocarcinoma in Situ (AIS), Invasive Cervical Carcinoma, high-grade Vulvar Intraepithelial Neoplasia (VIN 2/3), high-grade Vaginal Intraepithelial Neoplasia (VaIN 2/3), high-grade Anal Intraepithelial Neoplasia (AIN 2/3), vulvar cancer, vaginal cancer and anal cancer post 3 doses of the investigational vaccine as determined by histopathologic examination among subjects, who are naïve (seronegative) to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain negative to the relevant HPV type(s) as determined by HPV-DNA test and without abnormal cervical biopsy result through Month 7 (composite end point)
The combined incidence of specific HPV types related persistent infections for no less than 12 months and related diseases | Up to 60th month after full immunization.
  The combined incidence of HPV types 6/11/16/18/31/33/45/52/58-related persistent infections for no less than 12 months as determined by testing samples from consecutive visits, and cervical, vulvar, vaginal and anal diseases among subjects, who are naïve (seronegative) to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain negative to the relevant HPV type(s) as determined by HPV-DNA test and without abnormal cervical biopsy result through Month 7.

SECONDARY OUTCOMES:
Overall incidence of adverse events post vaccination | 0-30 days after each immunization
  Overall incidence of adverse events post vaccination
Overall incidence of adverse reactions post vaccination | 0-30 days after each immunization
  Overall incidence of adverse reactions post vaccination
Incidence of adverse reactions by severity post vaccination | 0-30 days after each immunization
  Incidence of adverse reactions by severity post vaccination
Percentage of subjects with one or more injection-site or non-injection-site | 0-30 days after each immunization
  Percentage of subjects with one or more injection-site or non-injection-site
Incidence of adverse event/adverse reaction by sign/symptom post vaccination | 0-30 days after each immunization
  Incidence of adverse event/adverse reaction by sign/symptom post vaccination
Severity of adverse event/adverse reaction post vaccination | 0-30 days after each immunization
  Severity of adverse event/adverse reaction post vaccination
Incidence of adverse reactions post each vaccination | 0-30 days after each immunization
  Incidence of adverse reactions post each vaccination
Incidence of serious adverse events that occur during the observation period | Through study completion, an average of 5 years
  Incidence of serious adverse events that occur during the observation period
Follow up the information on Pregnancy events through the interview, telephone call, and Safety follow-up Diary Card (Questionnaire). | Through study completion, an average of 5 years
  Follow up the information on Pregnancy events through the interview, telephone call, and Safety follow-up Diary Card (Questionnaire).
Follow up the information on birth/infant outcomes through the interview, telephone call, and Safety follow-up Diary Card (Questionnaire). | Through study completion, an average of 5 years
  Follow up the information on birth/infant outcomes through the interview, telephone call, and Safety follow-up Diary Card (Questionnaire).
Incidence of HPV types 6/11/16/18/31/33/45/52/58-related persistent infections for no less than 6 months | Up to 60th month after the first immunization
  Incidence of HPV types 6/11/16/18/31/33/45/52/58-related persistent infections for no less than 6 months as determined by testing samples from consecutive visits among subjects, who are naïve (seronegative) to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain negative to the relevant HPV type(s) as determined by HPV-DNA test and without abnormal cervical biopsy result through Month 7
GMTs of neutralizing antibody responses to vaccine HPV types determined among subjects who are seronegative | 7th month after the first immunization
  GMTs of neutralizing antibody responses and seroconversion rates to vaccine HPV types, as determined by Pseudovirus-based Neutralization Assay at week 4 post dose 3 in subjects who are naïve (seronegative) to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain negative to the relevant HPV type(s) as determined by HPV-DNA test and without abnormal cervical biopsy result through Month 7
Seroconversion rates to vaccine HPV types determined among subjects who are seronegative | 7th month after the first immunization
  Seroconversion rates to vaccine HPV types, as determined by Pseudovirus-based Neutralization Assay at week 4 post dose 3 in subjects who are naïve (seronegative) to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain negative to the relevant HPV type(s) as determined by HPV-DNA test and without abnormal cervical biopsy result through Month 7
The immune responses to HPV 6, 11, 16, 18, 31, 33, 45, 52 and 58, and their persistence in terms of GMTs of vaccine HPV type-specific neutralizing antibodies among the group who are seronegative | Up to the 60 months after the first immunization
  To evaluate immune responses to HPV 6, 11, 16, 18, 31, 33, 45, 52 and 58, and their persistence in terms of GMTs of vaccine HPV type-specific neutralizing antibodies, as determined by Pseudovirus-based Neutralization Assay , respectively among the group who are seronegative to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain
The immune responses to HPV 6, 11, 16, 18, 31, 33, 45, 52 and 58, and their persistence in terms of GMTs of vaccine HPV type-specific IgG antibodies among the group who are seronegative | Up to the 60 months after the first immunization
  To evaluate immune responses to HPV 6, 11, 16, 18, 31, 33, 45, 52 and 58, and their persistence in terms of GMTs of vaccine HPV type-specific IgG antibodies, as determined by ELISA assay, respectively among the group who are seronegative to the relevant HPV type(s) (HPV 6/11/16/18/31/33/45/52/58) at baseline and remain

CONTACTS AND LOCATIONS:
Overall Officials: Yongjiang Liu, Bachelor, Study Chair — Beijing Health Guard Biotechnology, Inc
Locations (3):
- China (3):
  - CDC, Guangdong Provinc, Guangzhou, Guangdong
  - CDC, Jiangsu Province, Nanjing, Jiangsu
  - CDC, Shanxi Province, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No
No informed consent was obtained to disclose the subject's data and sample test results.